CLINICAL TRIAL: NCT04554446
Title: The Effectiveness and Safety of T-MSAT on Inpatients With Acute Low Back Pain Caused by Traffic Accidents : A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2020-10
Record Dates: First submitted 2020-09-07; First posted 2020-09-18 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Low Back Pain; Medicine, Korean Traditional
Keywords: acupuncture therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-MSAT(Motion style acupuncture treatment using Traction) (Experimental): T-MSAT group receives 3 sessions of T-MSAT; on 2nd, 3rd, 4th day after hospitalization. A trained doctor of Korean medicine with clinical experience conducted the T-MSAT. And T-MSAT group is also treated with other Korean integrative medicine treatment everyday: acupuncture, chuna, pharmacoacupuncture and Korean herbal medicine.
  Interventions: Procedure: T-MSAT(Motion style acupuncture treatment using traction); Procedure: Korean medicine treatment
- Korean medicine treatment (Active Comparator): The control group is received Korean integrative medicine treatment everyday; acupuncture, chuna, pharmacoacupuncture and Korean herbal medicine.
  Interventions: Procedure: Korean medicine treatment

INTERVENTIONS:
Procedure: T-MSAT(Motion style acupuncture treatment using traction) — Motion Style Acupuncture Treatment(MSAT) is a therapeutic technique using acupuncture needle created in Jaseng Hospital. T-MSAT(Motion style acupuncture treatment using traction) is a kind of MSATs, and a treatment that improves musculoskeletal problems by pulling the patient's body through the device and giving instructions for walking while being acupuncture.
  Arms: T-MSAT(Motion style acupuncture treatment using Traction)
Procedure: Korean medicine treatment — acupuncture, chuna, pharmacoacupuncture and Korean herbal medicine.

SUMMARY:
This study is a single blind, randomized controlled trial. condition/disease: acute low-back pain treatment/intervention: Motion Style Acupuncture Treatment using Traction (T-MSAT)

DETAILED DESCRIPTION:
Motion Style Acupuncture Treatment(MSAT) is a therapeutic technique using acupuncture needle created in Jaseng Hospital. T-MSAT(Motion style acupuncture treatment using traction) is a kind of MSATs, and a treatment that improves musculoskeletal problems by pulling the patient's body through the device and giving instructions for walking while being acupuncture.This treatment involves patients with musculoskeletal pain to move the part of their body actively during acupuncture treatment under physicians' observation. This treatment is known to relieve pain and improve musculoskeletal disfunctions. However, there has been no specific studies for the effect of this treatment.

So, investigators conduct a randomized controlled trials to verify the effectiveness and safety of T-MSAT. From September 2020 to March 2021, investigators recruit 100 inpatients who are suffered from acute low-back pain with the numeric rating scale(NRS) over 5 by traffic accident(TA). For experimental group(n=50), investigators conduct T-MSAT three times(on 2nd, 3rd and 4th day of hospitalization) and other Korean medical treatment. For control group(n=50), just Korean medical treatment except T-MSAT is conducted. For these two groups, investigators compare NRS(Numeric Rating Scale), Visual Analogue Scale(VAS), Range Of Motion(ROM), , Oswestry Disability Index(ODI), the 12-Item Short Form Health Survey(SF-12), and PTSD Checklist for DSM(Diagnostic and Statistical Manual of Mental Disorders, DSM)-5(PCL-5)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19-70 years on the date they sign the consent form
* Patients with NRS ≥ 5 for low-back pain
* Patients who needs hospitalization due to acute low-back pain that occurred within 7 days after traffic accident
* Patients who provide consent to participate in the trial and return the informed consent form

Exclusion Criteria:

* Patients with a specific serious disease that may cause acute low-back pain: malignancy, fracture of lumbar spine, etc.
* Patients with progressive neurological deficits or with severe neurological symptoms
* The cause of pain is due to soft tissue disease, not the spine: tumors, fibromyalgia, rheumatoid arthritis, gout, etc.
* Patients with other chronic conditions that may interfere with the interpretation of the therapeutic effects or results: cardiovascular disease, kidney disease, diabetic neuropathy, dementia, epilepsy, etc.
* Patients who are difficult to walk due to leg disorder unrelated to low-back pain
* Patients who are taking steroids, immunosuppressants, mental illness drugs, or other drugs that may affect the results of the study
* Patients who are pregnant, planning to become pregnant, or are breastfeeding
* Patients who have had surgery or procedures of lumbar spine within the last three weeks
* Patients with a serious mental illness
* Patients who are participated in clinical trials other than observational studies without therapeutic intervention.
* Patients who are difficult to complete the research participation agreement
* Other patients whose participation in the trial is judged by a researcher to be problematic

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale(NRS) of low-back pain | Change from baseline VAS at 4 days
  The extent of acute low-back pain and discomfort was assessed using NRS. NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participants are asked to report their low-back pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.

SECONDARY OUTCOMES:
Numeric Rating Scale(NRS) of low-back pain | baseline(day1), day2, day3, day4, day of Discharge(up to 14days), week 12
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participants are asked to report their low-back pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
Visual Analogue Scale (VAS) of low-back pain | Baseline, day3, day4, day of discharge(up to 14days)
  VAS is an assessment index in which the patient records their pain on a 100mm line from 'no pain' at one end, and 'the most severe pain imaginable' at the other end.
Visual Analogue Scale (VAS) of leg pain | Baseline, day3, day4, day of discharge(up to 14days)
  VAS is an assessment index in which the patient records their pain on a 100mm line from 'no pain' at one end, and 'the most severe pain imaginable' at the other end.
Numeric Rating Scale(NRS) of leg pain | Baseline, day3, day4, day of discharge(up to 14days), week12
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10.
Range of movement (ROM) of flexion | Baseline, day3, day4, day of discharge(up to 14days)
  Range of movement (ROM) of flexion is measured.
Range of movement (ROM) of extension | Baseline, day3, day4, day of discharge(up to 14days)
  Range of movement (ROM) of extension is measured.
Range of movement (ROM) of left lateral flexion | Baseline, day3, day4, day of discharge(up to 14days)
  Range of movement (ROM) of left lateral flexion is measured.
Range of movement (ROM) of right lateral flexion | Baseline, day3, day4, day of discharge(up to 14days)
  Range of movement (ROM) of right lateral flexion is measured.
Range of movement (ROM) of left rotation | Baseline, day3, day4, day of discharge(up to 14days)
  Range of movement (ROM) of left rotation is measured.
Range of movement (ROM) of right rotation | Baseline, day3, day4, day of discharge(up to 14days)
  Range of movement (ROM) of right rotation is measured.
Oswestry Disability Index (ODI) | Baseline, day4, day of discharge(up to 14days), week12
  Functional disability questionnaire. The possible range of each item score is 0 to 5. Total score range: 0 (better outcome) to 100 (worse outcome)
Korean version of The Posttraumatic Stress Disorder Checklist for DSM-5(PCL-5-K) | Baseline, day4, day of discharge(up to 14days), week12
  The PCL-5(The Posttraumatic Stress Disorder Checklist for DSM-5) is a 20-item, 5-point-Likert-scale, self-report questionnaire to measure the PTSD symptoms in the DSM-536 and to diagnose PTSD. A higher score (out of 80) indicates severe PTSD.
12-item Short-Form Health Survey (SF-12) | Baseline, day4, day of discharge(up to 14days), week12
  The SF-12 is a shortened version of the Short Form-36 Health Survey (SF-36), which is a widely used instrument to assess health-related quality of life. The SF-12 consists of 12 questions across 8 domains, and higher scores indicate better health-related quality of life.
Patient Global Impression of Change (PGIC) | day4, day of discharge(up to 14days), week12
  The PGIC is an index that assesses improvements in functional limitation caused by whiplash injury. Participants rate the improvement in functional limitations after treatment on a 7-point Likert scale (1=Very much improved, 4=No change, 7=Very much worse). This index was originally developed for use in Psychology, but is currently used in various other medical fields to assess improvements in pain.
Drug Consumption | Baseline, day3, day4, day of discharge(up to 14days), week12 (every visit)
  Drug type and dose of prescribe for medicine, and type and frequency of other treatments
Adverse events | Baseline, day3, day4, day of discharge(up to 14days), week12 (every visit)
  Safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Dr., Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No